CLINICAL TRIAL: NCT02859857
Title: Phase 1, Dose-Escalation, Open-label, Safety and Pharmacokinetic, First in Human Study of BXQ-350 Administered as a Single Agent by Intravenous Infusion in Adult Patients With Advanced Solid Tumors and Recurrent High-Grade Gliomas
Brief Title: Phase 1 Study of BXQ-350 in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bexion Pharmaceuticals, Inc. (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BXQ-350.AA
Record Dates: First submitted 2016-07-29; First posted 2016-08-09 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Neoplasms
Keywords: Glioblastoma Multiforme; Solid Tumors; Ependymoma
MeSH Terms: conditions — Neoplasms; Glioblastoma; Ependymoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Rising dose; safety and tolerance (Experimental): Sequential cohorts of patients with advanced solid tumors and recurrent high-grade gliomas will be be treated with escalating doses of BXQ-350 until the MTD is established, or in the absence of a MAD, the highest planned DL is reached.
  Interventions: Drug: BXQ-350
- Solid tumor patients (Experimental): Cohort of patients with advanced solid tumors administered BXQ-350 at the MTD determined in Part 1 or at the highest planned DL if the MAD is not reached.
  Interventions: Drug: BXQ-350
- Glioblastoma Multiforme patients (Experimental): Cohort of patients with recurrent high-grade gliomas administered BXQ-350 at the MTD determined in Part 1 or at the highest planned DL if the MAD is not reached.
  Interventions: Drug: BXQ-350
- Gastrointestinal tumor patients (Experimental): Cohort of patients with Gastrointestinal tumors as defined in the protocol and administered BXQ-350 at the 2.4 mg/kg dose level.
  Interventions: Drug: BXQ-350
- Ependymoma tumor patients (Experimental): Cohort of patients with ependymoma administered BXQ-350 at the 2.4 mg/kg dose level.
  Interventions: Drug: BXQ-350
- Solid tumor patients other than HGG (Experimental): Cohort of patients with advanced solid tumors other than HGG administered BXQ-350 at the 2.4 mg/kg dose level.
  Interventions: Drug: BXQ-350

INTERVENTIONS:
Drug: BXQ-350 — BXQ-350 is a novel anti-neoplastic therapeutic agent configured from two components: Saposin C (SapC), an expressed (human) lysosomal protein, and the phospholipid dioleoylphosphatidyl-serine (DOPS), a phospholipid located on cell membranes. When both the components are assembled together stable SapC-DOPS nanovesicles are formed(clinical formulation BXQ-350).
  Other Names: SapC-DOPS

SUMMARY:
The objective of this study is to characterize the safety profile and determine the maximum tolerate dose (MTD) of BXQ-350, when given as a single agent at escalating doses, according to the investigational product (IP) related dose-limiting toxicities (DLTs) in patients with advanced solid tumors. Secondarily to assess the preliminary antitumor activity of BXQ-350 in solid tumors and recurrent high grade gliomas.

DETAILED DESCRIPTION:
This is a first in man study of BXQ-350, a novel anti-neoplastic therapeutic agent composed of two components: Saposin C (SapC), an expressed (human) lysosomal protein, and the phospholipid dioleoylphosphatidyl-serine (DOPS), a phospholipid located on cell membranes. When both the components are assembled together forming stable SapC-DOPS nanovesicles (clinical formulation BXQ-350), the agent exhibits the propensity to enter the body and brain, target cells in the tumor mass, and induce cell death.

The study is divided into 3 parts:

1. Dose Escalation Scheme Sequential cohorts of adult patients with advanced solid tumors and recurrent high-grade gliomas will be treated with escalating doses of BXQ-350 until the MTD is established, or in the absence of a MAD, the highest planned DL.
2. During Part 2, patients with advanced solid tumors and recurrent high-grade gliomas will be enrolled and administered BXQ-350 at the MTD determined in Part 1 or at the highest planned DL, if the MAD is not reached.
3. During Part 3, patients with either ependymoma, GI tumors , or advanced solid tumors other than HGG, will be enrolled and administered BXQ-350 at the 2.4 mg/kg dose level.

ELIGIBILITY:
Inclusion Criteria:

* Each patient must meet the following criteria:

  1. Provide signed, written informed consent prior to the initiation of any study-specific procedures
  2. Have histologically or cytologically confirmed diagnosis of advanced solid tumor cancer (excluding lymphomas) for which there is no further standard therapy or when standard therapy is contraindicated. Patients with HGG must have shown unequivocal evidence for recurrence or progression by MRI scan or must have histologically proven tumor recurrence.
  3. Patients with HGG: Have previously received radiotherapy and temozolomide
  4. For patients with HGG and receiving glucocorticoid therapy, must be on stable or decreasing equivalent daily dose of glucocorticoids for 2 weeks (14 days) prior to dose assignment
  5. Have measurable or non-measurable disease per RECIST 1.1 criteria for solid tumors and RANO criteria for HGG
  6. Are males or females aged ≥ 18 years
  7. Have Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 - 2
  8. Have acceptable liver function defined as:

     * Total serum bilirubin ≤ 1.5 × upper limit of normal for the study site (ULN) (in patients with known Gilbert Syndrome, total bilirubin ≤ 3 × ULN, with direct bilirubin ≤ 1.5 × ULN)
     * Aspartate Transaminase (AST), Serum Glutamic Oxaloacetic Transaminase (SGOT), Alanine Transaminase (ALT), Serum Glutamic-Pyruvic Transamine (SGPT) ≤ 3 × ULN (if liver metastases are present, then ≤ 5 × ULN is allowed)
     * Serum albumin ≥ 3 g/dL
  9. Have acceptable renal function defined as:

     Serum creatinine ≤ 1.5 × ULN, OR calculated creatinine clearance ≥ 45 mL/min for patients with creatinine levels above 1.5 mg/dL
  10. Have acceptable bone marrow function defined as:

      * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
      * Platelet count ≥ 100,000 cells/mm3
      * Hemoglobin > 9.0 g/dL
  11. Have acceptable coagulation parameters defined as:

      * International normalized ratio (INR) ≤ 2 × ULN
      * Activated partial thromboplastin time (aPTT) within normal limits
  12. Have a negative serum pregnancy test result at screening (for females of child bearing potential (FCBP); not applicable to patients who are unable to become pregnant, including those with tubal ligation, bilateral oophorectomy and/or hysterectomy, post-menopausal is defined as > 12 months since last menstrual cycle)
  13. FCBP and male patients whose sexual partner(s) are FCBP must agree to abstain from heterosexual activity or use a double barrier method of contraception (e.g., condom and occlusive cap with spermicide) or highly effective contraception (intrauterine device or system, established hormonal contraceptive methods on a stable dose from the time of the last menstrual cycle, or vasectomized partner with confirmed azoospermia) from the time of study entry to 1 month after the last day of treatment

Exclusion Criteria:

* Patients must not meet any of the following criteria:

  1. Have a concurrent malignancy or have had another malignancy within 1 year prior to initiation of screening (with the exception of adequately treated basal or squamous cell carcinoma, melanoma in situ, early-stage prostate cancer (T1a-cN0M0), ductal carcinoma in situ of the breast or cervical carcinoma in situ)
  2. Patients with solid tumors: Have received anticancer therapies, including radiation therapy, cytotoxic agents, targeted agents or endocrine therapy within 2 weeks prior to dose assignment
  3. Patients with HGG: Have received anticancer therapies including: radiation therapy to current site of disease within 12 weeks of dose assignment, targeted agent therapy within 2 weeks of dose assignment, nitrosoureas within 6 weeks of dose assignment, procarbazine within 3 weeks of dose assignment, or other cytotoxic agents within 4 weeks of dose assignment
  4. Have not recovered from toxicity of prior therapy defined as a return to < grade 1 at the time of dose assignment, graded according to CTCAE v4.03 (excluding alopecia, neuropathy, and lymphopenia)
  5. Have received prior treatment with any investigational drug within 4 weeks prior to dose assignment
  6. Have had major surgery other than a minor outpatient procedure within 4 weeks prior to dose assignment or have not recovered from major side effects of the surgery if more than 4 weeks have elapsed since surgery
  7. Have a history of cardiac dysfunction including:

     * Myocardial infarction within 6 months prior to initiation of screening
     * History of documented congestive heart failure (New York Heart Association functional classification III-IV) within 6 months prior to initiation of screening
     * Active cardiomyopathy
     * ECG with correctd QT interval (QTc) >450 msec in males or >470 msec in females at screening
  8. Have a known history of HIV seropositivity
  9. Are pregnant or nursing (lactating), where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive serum human chorionic gonadotropin (hCG) laboratory test
  10. Have symptomatic brain metastases or leptomeningeal disease
  11. Have active (acute or chronic) or uncontrolled severe infections
  12. Have active poor wound healing (delayed healing, wound infection or fistula)
  13. Have poorly controlled hypertension defined as blood pressure >160/90 on at least 2 repeated determinations on separate days within 2 weeks (14 days) prior to initiation of screening
  14. Have evidence of active clinically significant bleed (e.g., gastrointestinal bleed, hemoptysis, or gross hematuria) at screening
  15. Have other concurrent severe and/or uncontrolled medical condition that would, in the site Investigator's judgment contraindicate the patient's participation in the clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Part 1-MTD | 12 months
  · To determine the maximum tolerate dose (MTD) of BXQ-350, when given as a single agent at escalating doses, according to the investigational product (IP) related dose-limiting toxicities (DLTs) in patients with advanced solid tumors
Part 2-RECIST | 12 months
  ·To assess preliminary antitumor activity, defined as maximal radiological response during treatment using Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 (v1.1) criteria for solid tumors.
Part 2-RANO | 12 months
  To assess preliminary antitumor activity, defined as maximal radiological response during treatment Revised Assessment in Neuro-Oncology (RANO) criteria for recurrent high grade glioma (HGG), of BXQ-350 given as a single agent at the MTD, or highest planned dose level (DL), in the absence of a Maximum Administered Dose (MAD).
Part 3 - RECIST | 12 months
  To assess preliminary antitumor activity, defined as maximal radiological response during treatment using Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 (v1.1) criteria for solid tumors

SECONDARY OUTCOMES:
Part 2- Area under Curve (AUC) | 12 months
  ·To evaluate the AUC of BXQ-350
Part 2-Cmax | 12 months
  To evaluate the Cmax of BXQ-350
Part 2-half life | 12 months
  To evaluate the half-life (t1/2) of BXQ-350
Part 2-CL | 12 months
  To evaluate the clearance (CL) of BXQ-350
Part 2-Progression-free survival (PFS-6) | 12 months
  To evaluate progression free survival at 6 months
Part 2-time to response | 12 months
  To evaluate time to response
Part 2-duration of response | 12 months
  To evaluate duration of response

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of Cincinnati Barrett Center, Cincinnati, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No